CLINICAL TRIAL: NCT02131727
Title: The Kent State-Cuyahoga County Health Promotion Study
Brief Title: Hand Hygiene Randomized Cluster Intervention to Reduce Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: GoJo Industries, Akron OH (Unknown); Cuyahoga County Government Center (Unknown)
Responsible Party: Principal Investigator, Maggie Stedman-Smith, Assistant Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-050
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Respiratory Tract Infections; Gastrointestinal Infections
Keywords: hand hygiene; communicable diseases; respiratory tract infections; primary prevention; employees
MeSH Terms: conditions — Respiratory Tract Infections; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hand Hygiene Improvement Intervention (Experimental): Hand Hygiene Improvement Intervention: Participants receive a 4 minute training video about actions to take to reduce risk of respiratory and GI infections that includes hand hygiene practices, along with educational posters and hand hygiene supplies.
  Interventions: Behavioral: Hand Hygiene Improvement Intervention
- Ask Me 3 (Placebo Comparator): Participants in the control group received a 4 minute training video about the Ask Me 3 program for clearer communication with health care providers, a brochure, and a key chain containing principles for clear communication with health care providers.
  Interventions: Behavioral: Ask Me 3

INTERVENTIONS:
Behavioral: Hand Hygiene Improvement Intervention — Participants received a 4 minute video about protective hand hygiene behaviors and other activities (cough ettiquette, and staying home when ill) to reduce the risk of contracting respiratory tract and GI infections. In addition, motivational posters and hand hygiene supplies were distributed in the work setting.
  Arms: Hand Hygiene Improvement Intervention
Behavioral: Ask Me 3 — Participants in the control group received a 4 minute training video about the "Ask Me 3" program to promote effective communication with health care providers, along with an "Ask Me 3" brochure and a key-chain with the "Ask Me 3" principles for effective communication with health care providers.
  Arms: Ask Me 3

SUMMARY:
The purpose of this study is to determine if a simple intervention to improve hand hygiene, consisting of a 3-4 minute training video, on-site posters, and hand hygiene supplies, can reduce respiratory and GI illness among employees.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a simple random cluster intervention trial to improve hand hygiene, consisting of a 3-4 minute training video, on-site posters, and hand hygiene supplies, can reduce respiratory and GI illness among those in the intervention group compared to the control group. The intervention was performed among employees in a Midwestern public government setting. Employees in the treatment group received a 3-4 minute training video online that was embedded in the baseline survey. Motivational posters from the USDHHS encouraging proper hand hygiene were installed in the workplace, along with hand hygiene supplies. The control group received a program called "Ask Me 3" developed by the National Patient Safety Foundation; the intervention consisted of a 3-4 minute training video to encourage clear communication with their health care providers, a brochure discussing the Ask Me 3 principles of clear communication with health care providers, and a key-ring with the Ask Me 3 communication principles to promote more effective communication with health care providers at visits out side of work. The groups were followed monthly through surveys over the Internet for an average of three months after baseline to determine if a relative reduction in self-reported respiratory / GI infections occurred in the intervention group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* All employees in respective departments participating in this study were included in the inclusion criteria

Exclusion Criteria:

* No employees were excluded if they worked in the participating departments in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Relative reduction in self-reported respiratory and gastrointestinal infections | prior 30 days as elicited by self-report on four monthly surveys
  Monthly surveys elicited information among employees in both the intervention and the control group about self-reported usual hand hygiene practices, symptoms of respiratory and GI infections and missed work days due to these symptoms during the prior 30 days. After the close of the study, statistical analysis was conducted to determine relative reductions in the intervention group compared to the control group regarding: self-reported infections and work days missed due to such infections.
Self-reported missed days of work due to symptoms of respiratory and gastrointestinal (GI) infections | Monthly surveys for an average of three months
  Monthly surveys were administered over the Internet for an average of three months to determine if a relative reduction occurred in the intervention group compared to the control group in self-reported missed days from work due to symptoms of respiratory or GI infections.

SECONDARY OUTCOMES:
Self-reported usual daily hand hygiene behaviors | Monthly self-report surveys for an average of three months from baseline
  Monthly surveys were administered for an average of three months to determine if a relative improvement from self-reported hand hygiene behaviors was seen in the intervention group compared to the control group, from baseline information.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Stedman-Smith, Ph.D., M.P.H., Principal Investigator — Kent State University
Locations (1):
- Kent State University, Kent, Ohio, United States